CLINICAL TRIAL: NCT04346251
Title: Correlation Analysis of Refraction and Biometric Parameters in Chinese Schoolchildren
Brief Title: Correlation Between Refraction and Biometric Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: CCPMOH2017-China-1101
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To document the refractive status of Chinese schoolchildren and evaluate the association between the degree of refraction and biometric parameters.

DETAILED DESCRIPTION:
In this study, we will analyze the refractive status of schoolchildren and compare the ocular biometrics, including spherical equivalent refraction (SER), pupil distance (PD), corneal curvature (CC), high order aberration (HOA), and central corneal thickness (CCT) between boys and girls. Additionally, we investigate the correlation between the SER in diopters and the other biometric parameters, including PD, CC, HOA, CCT, and body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren aged from 6 to 15 years

Exclusion Criteria:

* with previous histories of cataracts, keratitis, strabismus, or other visual impairments
* with history of previous eye surgery
* with unreliable auto-refraction values
* unwilling to participate

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Schoolchildren aged 6 to 15 years will be included in this cross-sectional study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
refractive error in diopters and biometric Parameters | up to 1 year
  Multiple regression analysis will be performed to evaluate the correlations between SER and the other biometric parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China